CLINICAL TRIAL: NCT01721850
Title: Evaluation of the Safety and Efficacy of New Infant Formula and Its Effects on the Gastrointestinal Tolerance (Crying Time) in Infantile Colic: a Double-blind, Randomized, Controlled Intervention Study
Brief Title: Evaluation of Safety and Efficacy of New Infant Formula in Infantile Colic
Acronym: Coco
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial insurance could not be prolonged any more and expired
Sponsor: HiPP GmbH & Co. Vertrieb KG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HiPP-505092
Record Dates: First submitted 2012-10-30; First posted 2012-11-06 (Estimated); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Infantile Colic
Keywords: infant nutrition, infantile colic
MeSH Terms: conditions — Colic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- control formula (Active Comparator): infants are fed a commercial stage 1 infant formula during the first 4 months of life, according to protocol
  Interventions: Other: control formula
- intervention formula 1 group (Experimental): infants are fed hydrolyzed infant formula containing pre- and probiotics during the first 4 months of life, according to protocol
  Interventions: Other: intervention formula 1
- intervention formula 2 group (Experimental): infants are fed hydrolyzed infant formula containing pre- and probiotics during the first 4 months of life, according to protocol
  Interventions: Other: intervention formula 2

INTERVENTIONS:
Other: control formula — commercial stage 1 infant formula
  Arms: control formula
Other: intervention formula 1 — infant formula with hydrolyzed protein (type I) and pre- and probiotics
  Arms: intervention formula 1 group
Other: intervention formula 2 — infant formula with hydrolyzed protein (type II) and pre- and probiotics
  Arms: intervention formula 2 group

SUMMARY:
The study is conducted to examine the safety and efficacy of a new infant formula and its effects on the gastrointestinal tolerance in infants suffering from colic.

Primary hypothesis to be tested is: an infant formula with optimized composition improves colicky symptoms compared to a standard formula.

ELIGIBILITY:
Inclusion Criteria:

* Healthy term infants
* Subjects appropriate for gestational age between 35 and 41 weeks
* Subjects between 15-60 days old
* Subjects with birth weight between 2500 and 4200 g and regular weight gain (≥150g / week)
* Diagnosis of infantile colic according to modified Wessel criteria (Crying episodes lasting 3 or more hours/day and occurring at least 3 days/week for at least 1 week)
* Subjects exclusively bottle-fed at study entrance
* Day care of the child only by mother/father
* Provide written informed consent in accordance with legal requirement

Exclusion Criteria:

* Neonatal problems (respiratory distress, asphyxia, Hypoglycaemia, sepsis, NEC)
* Clinical evidence of chronic illness or gastrointestinal disorders (GER, gastroenteritis)
* Assumption of any kind of medication (except vitamin D, vitamin K and fluoride prophylaxis) during the week before the beginning of the study and during the study period
* Subjects receiving formula for special medical purposes
* Exclusively breast-fed infants
* Feeding of supplemental Pro- and/or Prebiotics two weeks prior to inclusion
* Allergic diseases (manifest atopic dermatitis, cow's milk allergy)
* Participation in any other clinical intervention

Ages: 15 Days to 60 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 169 (Actual)
Dates: Start 2011-12 (Actual); Primary Completion 2019-04 (Actual); Study Completion 2019-04 (Actual)

PRIMARY OUTCOMES:
daily total crying time | 28 days
  evaluation of the difference in the average reduction of daily crying time after 28 days of intervention between treatment and control group

SECONDARY OUTCOMES:
growth parameters | 90 days
  determination of body weight, length, head circumference
tolerance evaluated by stool characteristics, gastrointestinal disorders and side effects | 28 days
  stool characteristics: frequency, consistency and color; gastrointestinal disorders: regurgitation, obstipation; side effects: vomiting, diarrhea, skin reactions
formula intake | 28 days
  evaluation of average daily drinking amount and formula acceptance
intestinal microbiota | 0-28 days
  evaluation of changes in the composition of the intestinal microbiota (Lactobacilli, Bifidobacteria, Coliforms) after intervention

CONTACTS AND LOCATIONS:
Overall Officials: Francesco Savino, Dr., Principal Investigator — Ospedale Infantile Regina Margherita, Dipartimento di Scienze Pediatriche e dell'Adolescenza.
Locations (13):
- Germany (3):
  - Pediatric Office, Düsseldorf
  - Pediatric Office, Kehl
  - Pediatric Office, Mülheim
- Italy (10):
  - Pediatric office, Alba, Piedmont
  - Pediatric office, Borgone, Piedmont
  - Pediatric office, Carmagnola, Piedmont
  - Pediatric Office, Condove, Piedmont
  - Pediatric office, Mondovì, Piedmont
  - Pediatric office, San Mauro Torinese, Piedmont
  - Pediatric office, Turin, Piedmont
  - Pediatric Office, Turin, Piedmont
  - Pediatric Office, Volpiano, Piedmont
  - Pediatric Office, Volvera, Piedmont